CLINICAL TRIAL: NCT02740452
Title: Ligamys Technique Versus Standard Technique for the Anterior Cruciate Ligament Rupture
Brief Title: Anterior Cruciate Ligament Rupture
Acronym: LIGAMYS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Société Mathys SA for sponsoring Ligamys Device (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU 0260
Record Dates: First submitted 2016-03-25; First posted 2016-04-15 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2021-06

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Rupture; Anterior Cruciate Ligament (ACL); Laxity knee; Instability knee
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Rupture

ARMS (2):
- Ligamys technique (Other): Ligamys technique (device) or standard technique
  Interventions: Device: ligamys technique
- standard technique (Other): Ligamys technique (device) or standard technique
  Interventions: Other: standard technique (anatomic reconstruction)

INTERVENTIONS:
Device: ligamys technique — Ligamys technique (device) or standard technique
  Arms: Ligamys technique
Other: standard technique (anatomic reconstruction) — Ligamys technique (device) or standard technique
  Arms: standard technique

SUMMARY:
The assess results of Anterior Cruciate Ligament (ACL) repair with the Ligamys® surgical technique versus standard technique.

The aim of the study is to compare (laxity, instability, and safety) these two types of treatment by using a prospective, randomised multicenter analysis.

DETAILED DESCRIPTION:
The treatment of acute ruptures of the anterior cruciate ligament is surgical in some cases with ligamentoplasty technique.

Contrary to the classic ligamentoplasty, the treatment with Ligamys consists of promoting heating of the ligament itself by controlling mechanical environment.

It allows a "dynamic" stabilization of the torn Anterior Cruciate Ligament with in the 3 weekly following traumatism. These techniques may improve the recovery process, proprioceptive results, decrease morbidity of transplant harvesting and faster for the patients. It's all these issues we would like to assess with a randomised multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 35 years
* Primary Anterior Cruciate Ligament rupture
* signed patient consent
* surgery 21 days or less after traumatism for Ligamys technique

Exclusion Criteria:

* infection of the operating site
* previous osseous disease
* pregnant or nursing woman.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Measuring anterior knee laxity with KT 1000 arthrometer | at 12 months

SECONDARY OUTCOMES:
Tegnér scores | at 12 months
Lysholm scores | at 12 months
IKDC score safety | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane DESCAMPS, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France